CLINICAL TRIAL: NCT07223476
Title: Treatment Landscape and Real-World Dosing Patterns With CDK4/6 Inhibitors for HR+/HER2- Advanced/Metastatic Breast Cancer in Portugal
Brief Title: Treatment Landscape and Real-World Dosing Patterns With CDK4/6 Inhibitors for Breast Cancer in Portugal
Acronym: PORTRAIT
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011APT03
Record Dates: First submitted 2025-10-29; First posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: Cyclin-dependent Kinase 4/6 Inhibitor; Real-world
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Ribociclib Treatment Group: HR+/HER2- a/mBC patients with at least 1 month of ribociclib treatment.
- Palbociclib Treatment Group: HR+/HER2- a/mBC patients with at least 1 month of palbociclib treatment.
- Abemaciclib Treatment Group: HR+/HER2- a/mBC patients with at least 1 month of abemaciclib treatment.

SUMMARY:
Assess and characterize the real-world cyclin-dependent kinase 4/6 inhibitor (CDKI) use in advanced/metastatic breast cancer (a/mBC), evaluate treatment persistence, and quantify CDKI dose adjustments in Portugal.

This study used secondary data from the IQVIA database that collects data from hospital drug consumption. The study included 16 public hospitals across Portugal, for which data on consumption of drugs used in hormone receptor positive/human epidermal growth factor receptor 2 negative (HR+/HER2-) a/mBC treatment was available. Patient selection was based on a set of criteria considering all patients with treatments in the a/mBC setting with use of at least one CDKI from November 2018 to May 2023.

ELIGIBILITY:
Inclusion criteria:

* Male and female patients of all ages.
* Patients with at least one CDKI consumption from November 2018 to May 2023.
* Patients with consumptions in Gynecology and Oncology specialties.

Exclusion criteria:

* Consumption patterns of target drugs that are not compatible with any known a/mBC treatment regimen.
* Patients in early stages of breast cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 1926 (Actual)
Dates: Start 2024-03-29 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Number of Patients Treated With a CDKI Between November 2018 and May 2023 | Up to approximately 4 years and 6 months
Median Treatment Duration | Up to approximately 4 years and 6 months
Median Time to Next Treatment (TTNT) | Up to approximately 4 years and 6 months
  TTNT was calculated considering the time between the start of one treatment line and the start of the next treatment line.
Number of Patients With Dose Reductions by Treatment Length per Line of Treatment | Up to approximately 4 years and 6 months
  Patients were categorized as having 0, 1, or 2 dose reductions over 0-6 months, 7-12 months, and 12 months or more of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States